CLINICAL TRIAL: NCT05490732
Title: Pharmacokinetic Population Modeling of Methadone in Patients Managed for Opioid Opioid Addiction
Brief Title: Pharmacokinetic Modeling of Methadone
Acronym: PKMETHAHOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21_0614
Record Dates: First submitted 2022-07-21; First posted 2022-08-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Toxicomania
Keywords: pharmacokinetics; methadone; microsampling; modeling
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeutic drug monitoring of methadone (Experimental): 6 samplings per subject: 3 venipunctures and 3 microsamplings
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Patient will be subjected to 3 blood sampling over 24hours. At H0, H4 and H12-24.
  For each one, one microsampling and one venipuncture
  Other Names: Volumetric absorptive microsampling

SUMMARY:
The management of patients with opioid addiction is a challenge insofar as many distractors or variability factors can interfere with the control of the addiction, whether they are psychological, psychiatric, environmental, pharmacokinetic or pharmacodynamic. Understanding this variability is potentially to be able to adjust a priori a dosage and to identify the factors of clinical response. Few population pharmacokinetic models exist for methadone and they generally concern the management of pain in palliative care patients or the management of opioid withdrawal syndrome in neonates. The hypothesis is therefore that the creation of such a model would make it possible to reduce patients' withdrawal periods, to set a target for plasma concentrations with a view to reducing dosages, and to empower the patient in his choice to monitor blood concentrations facilitated by a minimally invasive sampling device.

ELIGIBILITY:
Inclusion Criteria:

* Major patients on methadone on the same dosage for at least 7 days.
* Hospitalization for withdrawal in the addictology department of La Colombière or consultation within the unit for the treatment of drug addiction and dependence (Addictology Department).
* 24 hours monitoring is possible and accepted

Exclusion Criteria:

* Patients that cannot be sampled because of weakened veins
* Unable to received information about the study
* Exclusion period determined by previous study
* Adult protected by law or patient under guardianship
* Not affiliated to french social security system
* Not able to give written inform consent
* Pregnant or breastfeeding woman
* Underaged patients (under 18 years old)
* Patient under court protection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-23 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | 18 months
  To evaluate and estimate methadone/EDDP (metabolite) Cmax for patients treated for opioid addiction.

SECONDARY OUTCOMES:
C12h-24h concentration | 18 months
  To evaluate and estimate methadone/EDDP (metabolite) concentration between 12 and 24h post-administration for patients treated for opioid addiction.
Residual concentration (C0) | 18 months
  To evaluate and estimate residual methadone/EDDP (metabolite) concentration for patients treated for opioid addiction.

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Cazaubon, phD,pharmD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No